CLINICAL TRIAL: NCT00329836
Title: A Research Study to Examine Cutaneous Allodynia and Cluster Headache
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Stephen D. Silberstein, Professor of Neurology, Thomas Jefferson University
Other Study IDs: CA/CH/01
Record Dates: First submitted 2006-05-24; First posted 2006-05-25 (Estimated); Results first posted 2011-08-16 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with cluster headache: Subjects with both episodic and chronic cluster (as defined by the International Headache Society-IHS) were enrolled.
  Interventions: Other: There are no interventions in the observational study. The symptom of allodynia was measured.

INTERVENTIONS:
Other: There are no interventions in the observational study. The symptom of allodynia was measured. — No intervention. Description of allodynia testing appears elsewhere in this document

SUMMARY:
This is a research study examining cutaneous allodynia and cluster headaches. Cutaneous allodynia means the feeling of pain or unpleasant sensation when normally non-painful stimuli (e.g. light touch) are applied to the skin. Many studies have been performed looking at the presence of cutaneous allodynia in patients with migraines; however, few studies have examined it in cluster headache patients. There is still much to be learned about the brain and how it functions if the investigators are to understand the underlying causes of cluster headache. It is important to explore cutaneous allodynia in cluster headache as it may help guide physicians with the care of these individuals. Sixty patients will be screened for this study. Thomas Jefferson University is the only center enrolling patients in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-75, inclusive
* Diagnosis of cluster headache, episodic or chronic.
* Patients with episodic CH can be either in active cluster period or not.
* Ability to read and understand an informed consent form, where the study protocol is described.

Exclusion Criteria:

* Patients with abnormal sensory findings on examination, or any known neurological disease that may affect skin sensation (peripheral neuropathy, multiple sclerosis, stroke, etc).
* Patients who are cognitively impaired, as determined by investigator
* Patients with significant psychiatric disorder that may affect their understanding of the study protocol and/or their cooperation with the investigators.
* Patients who had taken an acute pain medication within 24 hours prior to allodynia testing.
* Patients with skin diseases that may cause abnormal skin sensation.
* Patients who had been treated with a nerve block in the 4 week period prior to allodynia testing
* Patients who had been treated with Botulinum neurotoxin within the 4 month period prior to allodynia testing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with cluster headache
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2006-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham A. Ashkenazi, M.D., Principal Investigator — Jefferson Headache Center/ thomas Jefferson University
Locations (1):
- Jefferson Headache Center/ Thomas Jefferson University, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with cluster headache recruited from Jefferson Headache Center office practice or community. First subject enrolled 7/5/05. Last subject enrolled 6/9/06.
Period: Overall Study
Arm/Group | Subjects With Cluster Headache
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects With Cluster Headache
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Allodynia in Subjects With Cluster Headache
Description: Allodynia (discomfort to normal sensation) was assessed by brushing at constant rate of 2 brushes/sec and pressure allodynia with Von Frei hairs. Outcome (discomfort) was measured on a 100 mm visual analogue scale.
Time Frame: Allodynia was assessed at the screening visit
Population: All enrolled subjects were analyzed
Measure: Number; unit: participants
Arm/Group | Subjects With Cluster Headache
Number analyzed (Participants) | 41
participants | 20

ADVERSE EVENTS:
Arm/Group | Subjects With Cluster Headache
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes